CLINICAL TRIAL: NCT06119672
Title: Evaluation of the Efficacy of Supplementary Probiotic Capsules With Topical Clobetasol Propionate 0.05% in the Treatment of Oral Lichen Planus
Brief Title: Efficacy of Probiotic Capsules With Topical Clobetasol Propionate in OLP Treatment
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: October 6 University (Other)
Collaborators: Cairo University (Other)
Responsible Party: Principal Investigator, Amira Abdelwhab, lecturer, October 6 University
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 311122
Record Dates: First submitted 2023-09-25; First posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Oral Lichen Planus
Keywords: oral lichen planus; probiotics; clobetasol probionate
MeSH Terms: conditions — Lichen Planus, Oral | interventions — Adrenal Cortex Hormones; Orabase

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- systemic probiotic (A) (Active Comparator): Systemic probiotic capsules will be given twice daily in addition to topical application of topical clobetasol in orabase twice daily
  Interventions: Drug: Probiotic Blend Oral capsules; Drug: Corticosteroids for Local Oral Treatment
- topical corticosteroid (B) (Active Comparator): topical clobetasol in orabse application will be given 4 times daily ( 3 times after meals and once before bed time) prophylactic topical antifungal will be given in the fourth week to prevent candidal infection
  Interventions: Drug: Corticosteroids for Local Oral Treatment

INTERVENTIONS:
Drug: Probiotic Blend Oral capsules — probtiotic bend oral tablets from biovia will be adminestrated containing 4 strains ( twice daily) in addition to topical clobetasol application twice daily
  Arms: systemic probiotic (A)
Drug: Corticosteroids for Local Oral Treatment — topical clobetasol probionate in orabase application 4 times daily
  Other Names: clobetasol probionate in orabase

SUMMARY:
Oral lichen planus patients who will meet inclusion criteria will be divided into 2 groups

-The intervention group (Group P): This group will be randomly allocated to take one capsule twice daily during meal time at morning and evening of probiotics complex obtained from Biovea for 4 -week study period. Moreover, patients in this group will be instructed to apply clobetasole propionate in orabase gel 2 times daily for 4 weeks. Patients will receive their supply of the gel and probiotics every 2 weeks. The control group (Group B): This group will be randomly allocated to apply clobetasol propionate in orabase gel 4 times daily after meal times and before sleeping for 4 weeks. At the 3rd week this group will be instructed to apply miconazole gel 4 times daily as a prophylaxis for two weeks.

Salivary sample collection: Unstimulated salivary sample was collected from all participants twice , once at baseline and another time after 4 weeks from the study period. Saliva was collected in graduated clear test tubes to be used in the evaluation of candidal counts before and after treatment .

Patient's visits was at baseline, 2 weeks and 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are diagnosed with symptomatic lichen planus whether bullous erosive or erythematous oral lichen planus.
* Male or female patient with age range between 20-75 years old were included.
* medically free individuals

Exclusion Criteria:

* the use of systemic antibiotics, corticosteroids or immunosuppressive agents within four weeks prior to enrollment in the study.
* Pregnant females
* patients with history of systemic disorder affecting the immune system
* active liver diseases and cancer
* allergy or intolerance to probiotics.
* any other oral lesions

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-10-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
size wound | 0 , 2 weeks and 4 weeks
  thongprasom scale
Pain in oral cavity | 0 , 2 weeks and 4 weeks
  Numerical rating scale (0-10) 0= minimal pain 10 unbearable pain

SECONDARY OUTCOMES:
candidal load assessment | 0 and 4 weeks
  culturing technique in CFU unit

CONTACTS AND LOCATIONS:
Overall Officials: yasmine kamal, lecturer, Principal Investigator — Cairo University
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol